CLINICAL TRIAL: NCT00916721
Title: Memory Reconsolidation Blockade as a Novel Intervention for Nicotine Dependence
Acronym: SCP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, A. Eden Evins, Director Center for Addiction Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2007P-001903; NIH grant 207610
Record Dates: First submitted 2009-06-05; First posted 2009-06-09 (Estimated); Results first posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Smoking Cessation
Keywords: Smoking cessation; propranolol; memory reconsolidation blockade; craving
MeSH Terms: conditions — Smoking Cessation | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propranolol (Active Comparator): propranolol
  Interventions: Drug: Propranolol
- Placebo (Placebo Comparator): sugar pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranolol — Visit 2 (first smoking-related memory reactivation session) the subject will be given 0.67 mg/kg (minimum 40 mg; maximum 80 mg) of short-acting propranolol (or placebo) rounded to the nearest 10 mg. Ninety minutes after this dose, if subject has tolerated the short-acting dose well, and if systolic blood pressure has not fallen by 10 mmHg or more to below 100 mmHg, the subject will be given oral long-acting propranolol 1 mg/kg (minimum 60 mg; maximum 120 mg) or placebo rounded to the nearest 20 mg. . If the subject tolerates the combination dose well, during treatment phase (from visit 7 to 12), both the short- and long-acting doses will be given together immediately prior to memory reactivation.
  Other Names: Inderal
  Arms: Propranolol
Drug: Placebo — Visit 2 (first smoking-related memory reactivation session) the subject will be given 0.67 mg/kg (minimum 40 mg; maximum 80 mg) of short-acting propranolol (or placebo) rounded to the nearest 10 mg. Ninety minutes after this dose, if subject has tolerated the short-acting dose well, and if systolic blood pressure has not fallen by 10 mmHg or more to below 100 mmHg, the subject will be given oral long-acting propranolol 1 mg/kg (minimum 60 mg; maximum 120 mg) or placebo rounded to the nearest 20 mg. . If the subject tolerates the combination dose well, during treatment phase (from visit 7 to 12), both the short- and long-acting doses will be given together immediately prior to memory reactivation.
  Arms: Placebo

SUMMARY:
Smoking is the leading cause of preventable morbidity and mortality in the US. While approximately 70% of smokers attempt to quit each year, only 5-15% maintain abstinence for 12 months, even with effective pharmacological and psychological interventions. Novel therapies are needed for smoking cessation and relapse prevention. Previous studies show that early post-cessation craving or urge to smoke is a powerful predictor of relapse. A current model of the pathogenesis of addiction maintains that a substance of abuse causes a marked increase release in phasic dopamine release, which in turn strengthens or increases the salience of the memory of the drug experience, leading to a powerful and persistent memory that is easily activated, leading to drug craving and often to drug use. This highly salient memory is also implicated in the physiological arousal associated with craving responses to smoking cues. This process is thought to be implicated in relapse to drug use after even long periods of abstinence. Recent animal research indicates that retrieval returns a consolidated memory such as those associated with drug craving, to a labile state from which it must be restabilized to persist in a process termed reconsolidation. If memories of drug-related experiences are labile when reactivated, this could represent a window of opportunity in which the memory of drug use that underlies drug craving can be influenced pharmacologically. Our hypothesis is that post-reactivation administration of the B-adrenergic blocker, propranolol, following retrieval of drug-associated memories will reduce the strength or salience of the memory by influencing reconsolidation, a process called memory reconsolidation blockade. In this study we will test the hypothesis that a single dose of propranolol given one hour prior to smoking-related cue exposure (post-reactivation treatment) will decrease psychophysiological responses to smoking cues one week later and will predict clinical response to an ensuing series of 6 post-reactivation treatments with script-driven imagery and propranolol. In order to do so, we propose to conduct a randomized, double-blind, placebo-controlled trial of post-reactivation treatment with propranolol in 50 adult smokers. Outcome measures will include in physiological responses to smoking-related cues after one and six post-reactivation treatments and smoking behavior during the treatment and during a 3-month follow-up period.

DETAILED DESCRIPTION:
SPECIFIC AIMS

1. To evaluate, in current smokers, the efficacy of a single dose of study medication given an hour prior to smoking-related cue exposure (post-reactivation treatment) on psychophysiological response to smoking cues one week later.
2. To evaluate, during the smoking cessation process, the clinical effect of study medication in an ensuing series of 6 post-reactivation treatments on psychophysiologic response to smoking cues measured one week after the last post-reactivation treatment.
3. To evaluate whether medication effect on psychophysiologic response during a single memory reactivation session with script-driven imagery will predict clinical response to an ensuing series of 6 post-reactivation treatments with script-driven imagery and study medication.
4. . To assess whether a single post-reactivation treatment or series of six post-reactivation treatments is associated with reduction in self-reported craving for cigarettes as assessed with the Tiffany QSU.
5. To assess whether a series of six post-reactivation treatments is associated with reduction in smoking as assessed with self-report of cigarettes smoked per day and expired air Carbon monoxide.

To achieve these aims, we will conduct a double-blind, randomized, placebo-controlled trial in a convenience sample of 50 smokers.

ELIGIBILITY:
Inclusion:

* Healthy smokers aged 18-65 who have smoked at least 10 cigarettes/day for the past 3 months

Exclusion:

* Age <18 or >65
* Systolic blood pressure <100 mm Hg;
* Medical condition that contraindicates the administration of propranolol, e.g., history of congestive heart failure, heart block, insulin-dependent diabetes, chronic bronchitis, emphysema, or asthma. With regard to asthma, because many persons who say they have had an asthma attack, especially as a child, may only have had hay fever, another allergy, or another non-asthmatic episode, a blanket exclusion criterion may be overly restrictive. Therefore, asthma attacks will only be exclusionary if they a.) occurred within the past ten years, b.) occurred at any time in life if induced by a B-blocker, or c.) are currently being treated, regardless of the date of last occurrence. Cardiological consultation will be obtained as necessary;
* Previous adverse reaction to, or non-compliance with, a B-blocker;
* Current use of medication that may involve potentially dangerous interactions with propranolol, including, other B-blockers, antiarrhythmics, or calcium channel blockers.
* Use of drugs of abuse other than nicotine or caffeine, such as opiates, marijuana, cocaine, or amphetamines, as determined by saliva or urine testing;
* Pregnancy (in women of child-bearing potential, a pregnancy test will be performed) or breast-feeding;
* Current PTSD, or psychotic, melancholic, or bipolar disorder
* Diagnosis of major depressive disorder in the past 6 months or HAM-D score >15 at screening
* Current participation in any additional nicotine dependence treatment.
* An urgent need to stop smoking: subjects who receive placebo may not achieve optimal smoking cessation results.
* Inability to understand the study's procedures, risks, and side effects, or to otherwise give informed consent for participation;
* Subject candidate does not understand English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2008-04; Primary Completion 2010-07 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A. Eden Evins, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital - Center For Addiction Medicine, Boston, Massachusetts, United States

REFERENCES:
- [Background] Lee JL, Everitt BJ, Thomas KL. Independent cellular processes for hippocampal memory consolidation and reconsolidation. Science. 2004 May 7;304(5672):839-43. doi: 10.1126/science.1095760. Epub 2004 Apr 8. PMID 15073322
- [Background] Alberini CM. Mechanisms of memory stabilization: are consolidation and reconsolidation similar or distinct processes? Trends Neurosci. 2005 Jan;28(1):51-6. doi: 10.1016/j.tins.2004.11.001. PMID 15626497
- [Background] Suzuki A, Josselyn SA, Frankland PW, Masushige S, Silva AJ, Kida S. Memory reconsolidation and extinction have distinct temporal and biochemical signatures. J Neurosci. 2004 May 19;24(20):4787-95. doi: 10.1523/JNEUROSCI.5491-03.2004. PMID 15152039
- [Background] McGaugh JL. The amygdala modulates the consolidation of memories of emotionally arousing experiences. Annu Rev Neurosci. 2004;27:1-28. doi: 10.1146/annurev.neuro.27.070203.144157. PMID 15217324
- [Background] Pitman RK, Sanders KM, Zusman RM, Healy AR, Cheema F, Lasko NB, Cahill L, Orr SP. Pilot study of secondary prevention of posttraumatic stress disorder with propranolol. Biol Psychiatry. 2002 Jan 15;51(2):189-92. doi: 10.1016/s0006-3223(01)01279-3. PMID 11822998
- [Background] Vaiva G, Ducrocq F, Jezequel K, Averland B, Lestavel P, Brunet A, Marmar CR. Immediate treatment with propranolol decreases posttraumatic stress disorder two months after trauma. Biol Psychiatry. 2003 Nov 1;54(9):947-9. doi: 10.1016/s0006-3223(03)00412-8. PMID 14573324
- [Background] Przybyslawski J, Roullet P, Sara SJ. Attenuation of emotional and nonemotional memories after their reactivation: role of beta adrenergic receptors. J Neurosci. 1999 Aug 1;19(15):6623-8. doi: 10.1523/JNEUROSCI.19-15-06623.1999. PMID 10414990
- [Background] Debiec J, Ledoux JE. Disruption of reconsolidation but not consolidation of auditory fear conditioning by noradrenergic blockade in the amygdala. Neuroscience. 2004;129(2):267-72. doi: 10.1016/j.neuroscience.2004.08.018. PMID 15501585
- [Background] Orr SP, Metzger LJ, Pitman RK. Psychophysiology of post-traumatic stress disorder. Psychiatr Clin North Am. 2002 Jun;25(2):271-93. doi: 10.1016/s0193-953x(01)00007-7. PMID 12136501
- [Background] Diergaarde L, Schoffelmeer AN, De Vries TJ. Beta-adrenoceptor mediated inhibition of long-term reward-related memory reconsolidation. Behav Brain Res. 2006 Jun 30;170(2):333-6. doi: 10.1016/j.bbr.2006.02.014. Epub 2006 Apr 5. PMID 16600394
- [Background] Bernardi RE, Lattal KM, Berger SP. Postretrieval propranolol disrupts a cocaine conditioned place preference. Neuroreport. 2006 Sep 18;17(13):1443-7. doi: 10.1097/01.wnr.0000233098.20655.26. PMID 16932155
- [Background] Robinson MJ, Franklin KB. Central but not peripheral beta-adrenergic antagonism blocks reconsolidation for a morphine place preference. Behav Brain Res. 2007 Aug 22;182(1):129-34. doi: 10.1016/j.bbr.2007.05.023. Epub 2007 May 24. PMID 17604134

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Treatment seeking adults smokers were enrolled from May 2008 to March 2010 at the Center for Addiction Medicine of the Massachusetts General Hospital, in compliance with the Declaration of Helsinki, the U.S. Food and Drug Administration guidelines, and the International Conference on Harmonization Good Clinical Practices Guidelines.
Pre-assignment Details: 39 were excluded before randomization: Did not meet inclusion criteria (21),Declined to participate (18) Three participants were discontinued before receiving study medication: due to bradycardia (1), cocaine use (1), recent use of albuterol (1)
Groups:
- Propranolol: A single oral dose of propranolol or identical placebo capsule in a double-blind fashion. Propranolol dose was 0.67 mg/kg of the short-acting formulation, rounded to the nearest 10 mg, with a minimum dose of 40 mg and a maximum dose of 80 mg
- Placebo: A single oral dose of identical placebo capsule in a double-blind fashion
Period: Overall Study
Arm/Group | Propranolol | Placebo
Started | 35 | 39
Completed | 25 | 29
Not Completed | 10 | 10
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 6 | 3
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Protocol Violation | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Propranolol | Placebo | Total
Number analyzed (Participants) | 35 | 39 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 39 | 74
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (10.9) | 42.5 (9.84) | 42.1 (10.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 20
  Male | 27 | 27 | 54
Region of Enrollment [Number; unit: participants]
  United States | 35 | 39 | 74

OUTCOME MEASURES:

1. Secondary Outcome: Change in Craving Level to Smoking Cues Caused by Smoking Cues, Measured Using Script Driven Imagery
Description: Craving level will be measured using a 8 point Visual Analogue Scale (VAS) of craving. Participants will be ask "How much do you want a cigarette right now" Participants will answer accordingly: 0=no desire at all; 7=unable to resist craving
Time Frame: Craving level was measured at visit 3, after presentation of two neutral and two smoking scripts
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 25 | 29
units on a scale | 5.52 (1.1) | 4.3 (2.1)

2. Primary Outcome: Change in the Skin Conductance Level, Caused by Smoking Cues, Measured Using Script Driven Imagery
Description: Skin conductance level was obtained through 9-mm (sensor diameter) Ag/AgCl electrodes filled with isotonic paste placed on the non-dominant hypothenar surface using a constant-voltage technique. A Coulbourn Modular Instrument System was used to measure SC during 4 periods; baseline, reading, imagery and recovery.
Time Frame: skin conductance was measured at visit 3, after presentation of two neutral and two smoking scripts
Measure: Mean (Standard Deviation); unit: µS
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 25 | 29
µS | 0.107 (0.728) | -0.040 (0.337)
Statistical Analysis 1: Comparison: Propranolol vs Placebo; Test type: Superiority or Other; p = 0.05, Mixed Models Analysis; Multiple significance testing:we adjusted p-value by controlling the expected proportion of falsely rejected hypotheses:false discovery rate,Benjamini

3. Primary Outcome: Change in Heart Rate (Beats Per Minute), Caused by Smoking Cues, Measured Using Script Driven Imagery
Description: Heart rate was measured through 9-mm (sensor diameter) Ag/AgCl electrodes filled with electrolytic paste and placed on the medial surface of each forearm. Amplified electrocardiogram signal will input to a tachometer that will provide a voltage output reflecting interbeat interval, which will be transformed to HR. A Coulbourn Modular Instrument System was used to measure HR during 4 periods; baseline, reading, imagery and recovery
Time Frame: Heart rate was measured at visit 3, after presentation of two neutral and two smoking scripts
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 25 | 29
beats per minute | 0.877 (2.285) | 1.162 (2.064)

4. Primary Outcome: Change in the Corrugator Muscle (EMG) Level, Caused by Smoking Cues, Measured Using Script Driven Imagery
Description: Corrugator EMG will be obtained through Ag/AgCl electrodes. The amplified EMG signal will be integrated using a 300-msec. time constant. A Coulbourn Modular Instrument System was used to measure corrugator EMG during 4 periods; baseline, reading, imagery and recovery
Time Frame: Corrugator EMG level was measured at visit 3, after presentation of two neutral and two smoking scripts
Measure: Mean (Standard Deviation); unit: µV
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 25 | 29
µV | 0.479 (1.309) | 1.464 (3.394)

ADVERSE EVENTS:
Arm/Group | Propranolol | Placebo
Serious Adverse Events (participants affected / at risk) | 1/35 | 0/39
Other Adverse Events (participants affected / at risk) | 6/35 | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propranolol (N=35) | Placebo (N=39)
major depressive episode and worsen anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propranolol (N=35) | Placebo (N=39)
bradycardia (Vascular disorders) | 6 (6) | 0 (0) — transient, asymptomatic bradycardia, i.e., HR< 50 beats per minute after taking short-acting propranolol.

LIMITATIONS AND CAVEATS:
Subjects were asked to not smoke for 12 hrs prior propranolol.Then were permitted to smoke throughout the week prior physiologic testing.Possibly each smoking experience presented a potential opportunity for the creation of new smoking memories.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No